CLINICAL TRIAL: NCT03598894
Title: Non-dipping Hypertension and the Human Chronobiome
Brief Title: Hypertension Chronobiome
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 828944
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Timed blood, saliva, swab, stool, urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case NDHT: Healthy non-dipping hypertensives 'NDHT' (24h mean wake SBP >145mmHg at baseline and a decline of <10% between mean day time and night time systolic pressures)
  Interventions: Other: Ambulatory blood pressure measurements
- Control NT: matched healthy normotensives 'NT' (24h mean wake SBP <120mmHg)
  Interventions: Other: Ambulatory blood pressure measurements
- Control DHT: matched dipping hypertensives 'DHT' (24h mean wake SBP >145mmHg and a decline of >10% between mean day time and night time systolic pressures)
  Interventions: Other: Ambulatory blood pressure measurements

INTERVENTIONS:
Other: Ambulatory blood pressure measurements — Blood pressure will be assessed with ambulatory blood pressure measurements over the course of a day to discern day/night differences

SUMMARY:
Hypertension is a common condition with a concomitant burden of stroke, kidney disease and myocardial infarction. Its prevalence in developed societies is increasing as they age, and in less developed countries, as their populations assume aspects of the Western diet and lifestyle. Nocturnal non-dipping hypertension (NDHT) - the failure of blood pressure (BP) to dip at night - is estimated to complicate ~40% of hypertensives and is associated with poor outcomes. Randomized controlled trials have shown that a reduction of daytime systolic blood pressure by as little as 5mmHg on average (towards a target of 140mmHg) translates into a measurable clinical benefit. The peak nocturnal difference may be ~15-20mmHg systolic, illustrating the substantial potential for incremental benefit by adequate blood pressure control across the 24 hour cycle in this population. In this study, the investigators wish (i) to establish through repeated assessment, the stability of the non-dipping phenotype (Phase 1), and (ii) to deeply phenotype non-dippers by using parameters assessing day/night patterns, the chronobiome (Phase 2). To facilitate data collection over the course of the study, the investigators use wearable devices and mobile phone applications.

ELIGIBILITY:
Phase 1: Inclusion Criteria (Stability of the non-dipping phenotype)

1. >18 years of age,
2. Upper arm with intact skin, i.e. without areas of breached or injured skin visible, for ABP measurements,
3. 24h mean wake SBP >145mmHg at baseline from 24hr-ABPM readings within the past 12 months,
4. Decline of <10% between mean day time and night time systolic pressures quantified per 24hr-ABPM within the past 6 months,
5. Own a smartphone.

Phase 1: Exclusion Criteria (Stability of the non-dipping phenotype)

1. Known history of severe psychiatric or cognitive conditions, for example mania, schizophrenia, or mental retardation.
2. Shift work, defined as recurring work between 22:00-05:00,
3. History of clinically significant obstructive sleep apnea;
4. Urine creatinine > 1.5 mg/dl in men or >1.3 mg/del in women,
5. Significant liver disease (>3x upper limit of normal),
6. Diabetes mellitus,
7. Transmeridian travel across ≥2 time zones in the month prior to ABP sessions,
8. Planned transmeridian travel across more than ≥2 time zones during the planned study activities;
9. > 2 drinks of alcohol per day;
10. Use of illicit drugs which affect blood pressure;
11. Use of pacemaker or implantable Cardioverter Defibrillator, (ICD);
12. Bilateral mastectomy;
13. Hypotension, defined as 90/60 mmHg assessed during the screening visit from ≥ 3 in-office measurements initiated after 10 minutes in seated upright position with 5 minute intervals between measurements;
14. History of Raynaud's phenomenon;
15. Known allergy against natural latex rubber (contained in ABP bladder and tubing);
16. Nursing or pregnant females.

Phase 2: Inclusion Criteria (Deeply phenotyping non-dipping hypertensives)

Inclusion Cohort 1 (case): non-dipping hypertensives 'NDHT'

1. >18 years of age,
2. Upper arm with intact skin, i.e. without areas of breached or injured skin visible, for ABP measurements,
3. 24h mean wake SBP >145mmHg from 24hr-ABPM readings confirmed per data base query within the past 12 months prior to enrollment into Phase 1 and across two subsequent 24hr-ABP sessions during Phase 1,
4. Decline of <10% between mean day time and night time systolic pressures from 24hr-ABPM readings confirmed per data base query within the past 12 months prior to enrollment into Phase 1 and across two subsequent 24hr-ABP sessions during Phase 1,
5. Own a smartphone.

Inclusion Cohort 2 (control): matched healthy normotensives 'NT'

1. >18 years of age,
2. Upper arm with intact skin, i.e. without areas of breached or injured skin visible, for ABP measurements,
3. Healthy (as assessed by health history, physical exam and screening lab work),
4. 24h mean wake SBP <130mmHg quantified per 24hr-ABPM,
5. Own a smartphone. 4.3.3 Inclusion Cohort 3 (control): matched dipping hypertensives 'DHT'

1) >18 years of age, 2) Upper arm with intact skin, i.e. without areas of breached or injured skin visible, for ABP measurements,

1. 24h mean wake SBP >145mmHg from 24hr-ABPM readings,
2. Decline of >10% between mean day time and night time systolic pressures from 24hr-ABPM readings,
3. Own a smartphone.

Phase 2 - Exclusion Criteria Cohorts 1-3

1. History of severe psychiatric illness or cognitive conditions, for example ( mania, schizophrenia, or mental retardation;
2. Shift work, defined as recurring work between 22:00-05:00;
3. Clinically significant obstructive sleep apnea as assessed per WatchPAT device;
4. Urine creatinine > 1.5 mg/dl in men or >1.3 mg/del in women;
5. Significant liver disease (>3x upper limit of normal);
6. Diabetes mellitus;
7. Past diagnosis of gastroesophageal reflux disease,
8. Transmeridian travel across ≥2 time zones in the two weeks before the 48hr deep phenotype sessions;
9. Frequent transmeridian flyer (≥2 flights per month) across more than ≥2 time zones during the 12 months of study activities;
10. Use of oral or intravenous antibiotics in the 6 months prior to enrollment;
11. Any contraindication listed below in the separate paragraph "Contraindications for the use of CorTemp® Disposable Temperature Sensors";
12. Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening;
13. > 2 drinks of alcohol per day;
14. Use of illicit drugs which affect blood pressure;
15. Nursing or pregnant (pregnancy will be repeatedly assessed at the beginning of each of the four inpatient visits, i.e. prior to the start of blood draws);
16. Use of pacemaker or implantable Cardioverter Defibrillator, (ICD)
17. Bilateral mastectomy;
18. Hypotension, defined as 90/60 mmHg assessed during the screening visit from ≥ 3 in-office measurements initiated after 10 minutes in seated upright position with 5 minute intervals between measurements;
19. History of Raynaud's phenomenon;
20. Known allergy against natural latex rubber (contained in ABP bladder and tubing);
21. Subjects taking medication with alpha-blockers;
22. History of clinically significant arrhythmias;
23. Subjects with a history of being particularly susceptible to vomiting or nausea;
24. BMI ≥ 30;
25. History of any type of GI Surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1 (case): Individuals with (Phase 1-) confirmed non-dipping phenotype 'NDHT'; Cohort 2 (control): matched healthy normotensives 'NT' (24h mean wake SBP <120mmHg); Cohort 3 (control): matched dipping hypertensives 'DHT' (24h mean wake SBP >145mmHg and a decline of >10% between mean day time and night time systolic pressures);
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure [mmHg] | 24-48 hours
  Ambulatory blood pressure measurements (ABPM)

SECONDARY OUTCOMES:
Dipping status [dimensionless ratio] | 24-48 hours
  Ratio of ambulatory blood pressure measurements during sleep and waking hours

CONTACTS AND LOCATIONS:
Overall Officials: Garret FitzGerald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
to be determined

REFERENCES:
- [Background] Skarke C, Lahens NF, Rhoades SD, Campbell A, Bittinger K, Bailey A, Hoffmann C, Olson RS, Chen L, Yang G, Price TS, Moore JH, Bushman FD, Greene CS, Grant GR, Weljie AM, FitzGerald GA. A Pilot Characterization of the Human Chronobiome. Sci Rep. 2017 Dec 7;7(1):17141. doi: 10.1038/s41598-017-17362-6. PMID 29215023